CLINICAL TRIAL: NCT01902719
Title: Family and Community Intervention to Address Hypertension Disparities
Brief Title: Achieving Blood Pressure Control Together Study
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00078591; 1P50HL105187 (NIH)
Record Dates: First submitted 2013-07-16; First posted 2013-07-18 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Community Health Workers; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Community Health Worker (CHW) Intervention (Experimental): Participants randomized to this arm will receive the Community Health Worker Intervention that will include training in the use of home blood pressure machine, education on diet and exercise, and one-on-one support to assist with overcoming barriers to hypertension control (e.g., accessing healthcare, social and community services).
  Interventions: Behavioral: Community Health Worker (CHW) Intervention
- CHW Intervention and Communication Skills Training (Experimental): Participants randomized to this arm will receive the Community Health Worker Intervention and a communication skills training to partner with their physician providers in a way that encourages their greater involvement and shared decision-making with their physicians about hypertension care.
  Interventions: Behavioral: Community Health Worker (CHW) Intervention; Behavioral: Communication Skills Training
- CHW and Problem Solving Skills Training (Experimental): Participants randomized to this arm will receive the Community Health Worker Intervention and the Problem Solving Skills Training Intervention, a 9-week peer based self-management intervention to help patients improve their hypertension self-management by learning and employing skills to overcome their self-identified barriers to self-management.
  Interventions: Behavioral: Community Health Worker (CHW) Intervention; Behavioral: Problem Solving Skills Training

INTERVENTIONS:
Behavioral: Community Health Worker (CHW) Intervention — Receipt of training in use of home blood pressure machine, education about diet, exercise and physical activities to lower blood pressure, and continued support from a trained community health worker.
Behavioral: Communication Skills Training — Receipt of "Do My PART" (P-Prepare for Visit, A- Act at visit, R-Review doctor's recommendations, T-Take home recommendations)communication skills training.
  Arms: CHW Intervention and Communication Skills Training
Behavioral: Problem Solving Skills Training — Receipt of a 9-week group based self-management intervention designed to help patients identify and solve self-identified barriers to hypertension control.
  Arms: CHW and Problem Solving Skills Training

SUMMARY:
African Americans represent a particularly vulnerable subgroup of persons with hypertension, as they are more likely than Whites to have hypertension, equally as likely to be aware of it and to be treated for it, but less likely to achieve blood pressure control while receiving treatment. African Americans are also more likely than Whites to suffer end organ damage as a result of hypertension. Patients' hypertension self-management behaviors (including adherence to prescribed care, self-blood pressure monitoring, lifestyle changes, and shared medical decision-making) represent a cornerstone of hypertension therapy. Evidence suggests some African Americans with hypertension may experience difficulties carrying out positive self-management behaviors, in part due to cultural beliefs and practices, knowledge and perceptions regarding the nature and consequences hypertension, and lack of systems to support ongoing engagement in prescribed care within their communities. Substantial evidence has demonstrated the important role of family and community support in improving patients' management of a variety of chronic illnesses.

The goal of this study is to rigorously test the effectiveness of hypertension self-management interventions that engage African American patients, their families, and their community-level resources to improve African American patients' blood pressure.

We hypothesize patients' hypertension control rates may be improved when combining community health worker self-management support with other types of hypertension self-management skills training.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* African American/Black
* English speaking
* Two Blood Pressure values >=140/>=90 in 6 months prior
* Seen at East Baltimore Medical Center

Exclusion Criteria:

* 18 years and less
* Non African American/Black
* Not English speaking
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Control | 12 months
  Hypertension control based on JNC-7 guidelines and changes in systolic and diastolic blood pressure. Blood pressure (BP) will be measured by trained and certified observers during regularly scheduled clinical visits at EBMC using an automatic oscillometric monitor (Omron HEM 907-XL). This device programs a five-minute delay before activation and has a 30-second delay between the triplicate measurements. We will use two measures - the average of all three measurements and the average of the last two measurements - obtained at each time point at baseline, 4 months, and 12 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh E Boulware, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins East Baltimore Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Murphy KA, Greer RC, Roter DL, Crews DC, Ephraim PL, Carson KA, Cooper LA, Albert MC, Boulware LE. Awareness and Discussions About Chronic Kidney Disease Among African-Americans with Chronic Kidney Disease and Hypertension: a Mixed Methods Study. J Gen Intern Med. 2020 Jan;35(1):298-306. doi: 10.1007/s11606-019-05540-3. Epub 2019 Nov 12. PMID 31720962
- [Derived] Boulware LE, Ephraim PL, Hill-Briggs F, Roter DL, Bone LR, Wolff JL, Lewis-Boyer L, Levine DM, Greer RC, Crews DC, Gudzune KA, Albert MC, Ramamurthi HC, Ameling JM, Davenport CA, Lee HJ, Pendergast JF, Wang NY, Carson KA, Sneed V, Gayles DJ, Flynn SJ, Monroe D, Hickman D, Purnell L, Simmons M, Fisher A, DePasquale N, Charleston J, Aboutamar HJ, Cabacungan AN, Cooper LA. Hypertension Self-management in Socially Disadvantaged African Americans: the Achieving Blood Pressure Control Together (ACT) Randomized Comparative Effectiveness Trial. J Gen Intern Med. 2020 Jan;35(1):142-152. doi: 10.1007/s11606-019-05396-7. Epub 2019 Nov 8. PMID 31705466